CLINICAL TRIAL: NCT05362877
Title: The Effect of Earplugs on Myogenous Temporomandibular Disorders
Brief Title: The Use of Earplugs on Temporomandibular Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr. Merve Benli, Assistant professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1302
Record Dates: First submitted 2022-01-25; First posted 2022-05-05 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Ear Protective Devices; Temporomandibular Joint Disorders; Physical Therapy Modalities
Keywords: Splints
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Ear Protective Devices; Occlusal Splints; Exercise

STUDY DESIGN:
Intervention Model Description: randomised controlled clinical trial
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Earplug (Experimental): Earplug group- using earplugs, n=20 Patients will use only earplugs
  Interventions: Device: Earplug
- Splint (Experimental): Occlusal splint group- using occlusal splints, n=20 Patients will use only occlusal splints
  Interventions: Device: occlusal splint
- Physical (Experimental): Exercise group- using physical therapy, n=20 Patients will do only exercise
  Interventions: Other: exercise
- control group (No Intervention): Control group-no intervention, n=20
- Earplug and splint (Experimental): Earplug group- using earplugs and splints, n=20 Patients will use both interventions
  Interventions: Device: Earplug; Device: occlusal splint
- Earplug and Physical (Experimental): Earplug group- using earplugs and exercise, n=20 Patients will use both interventions
  Interventions: Device: Earplug; Other: exercise

INTERVENTIONS:
Device: Earplug — Using earplugs to reduce the symptoms of temporomandibular disorder
  Arms: Earplug; Earplug and Physical; Earplug and splint
Device: occlusal splint — Using occlusal splints to reduce the symptoms of temporomandibular disorder
  Arms: Earplug and splint; Splint
Other: exercise — Applying exercise to reduce the symptoms of temporomandibular disorder
  Arms: Earplug and Physical; Physical

SUMMARY:
The term temporomandibular joint disorder (TMD) refers to a group of disorders affecting the temporomandibular joint and/or muscles of mastication. Typical symptoms are; joint noises, pain, and limited mouth opening. Many therapeutic modalities have been advocated for the treatment of TMD as intraoral splints, laser, ultrasound, physical therapy, surgery, and medications with inconsistent reported results due to the multifactorial etiology of this disorder. Although intraoral splints are the most widely used therapy, it has some drawbacks as being inconvenient for the patient due to their relatively large size interferes with eating and affects speech, therefore their use is mostly limited to sleeping time, which decreases its effectiveness.

Recently some commercial earplugs that claim to treat TMD have been introduced, however, there is no validated data regarding these appliances. Thus, this study aimss to evaluate the possible effect of earplugs on myogenous TMD.

ELIGIBILITY:
Inclusion Criteria:

* Pain in masticatory muscles for at least 3 months according to the DC/TMD
* Having a stable medication regimen for at least 1 month
* Age of 18-65 years
* Minimum pain intensity of 50 mm on a 100 mm visual analog scale (VAS)
* No concomitant systemic disease
* Natural posterior occlusion.

Exclusion Criteria:

* Undergoing physical therapy
* Using muscle relaxants and/or NSAIDs
* Previous TMD treatment more recently than one year
* Major psychosocial problems
* Undergoing orthodontic treatment
* Wearing removable prosthesis
* Pregnancy
* History of facial trauma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-12-03 (Actual)

PRIMARY OUTCOMES:
Values of maximal mouth opening(millimeter) | 2 months
  Evaluating mouth opening by using digital caliper

SECONDARY OUTCOMES:
Pain perception | 2 months
  Evaluating pain perception of the patients by using visual analogue scale and measuring pain response with self-evaluation and reporting (Minimum value: 0; maximum value:10)

OTHER OUTCOMES:
Symptom Severity | 2 months
  Evaluating temporomandibuler symptoms by using Symptom Severity Index

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul university,Faculty of Dentistry, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided